CLINICAL TRIAL: NCT06657547
Title: Urinary Concentration After Salmeterol in Well-trained Men and Females
Brief Title: Urinary Concentration After Salmeterol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Hostrup, PhD, Associate Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: SALM_urine
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: Urinary concentration; Beta2-adrenergic stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Normal conditions (Active Comparator): Urine samples collected after various performance tests in normal conditions
  Interventions: Other: Normal conditions
- Heated conditions (Experimental): Urine samples collected after various performance tests in heated conditions
  Interventions: Other: Heated conditions
- Salmeterol inhalation and urine samples (Other): Participants are administered daily salmeterol inhalation from an MDI device and are required to collect spot urine samples at home.
  Interventions: Drug: Salmeterol inhalation and urine samples

INTERVENTIONS:
Other: Normal conditions — Participants are administered salmeterol, after which they perform various performance tests in normal conditions. Following the administration of salmeterol, urine samples are collected over the next 24 hours at intervals of 0.5, 1, 2, 4, 8, and 24 hours after administration.
  Arms: Normal conditions
Other: Heated conditions — Participants are administered salmeterol, after which they perform various performance tests in heated conditions. Following the administration of salmeterol, urine samples are collected over the next 24 hours at intervals of 0.5, 1, 2, 4, 8, and 24 hours after administration.
  Arms: Heated conditions
Drug: Salmeterol inhalation and urine samples — After the experimental day under normal conditions, all participants are administered 200 µg of salmeterol daily (8 puffs from the MDI device) during a 6-day intervention period. Two hours after inhalation, the participants collect spot urine samples at home
  Arms: Salmeterol inhalation and urine samples

SUMMARY:
The purpose of the project is to investigate urine concentration after inhalation of salmeterol. This will be examined following acute physical activity under both normal conditions and heated conditions.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* Age 18-40
* Physically active >5 hours a week
* Maximum oxygen uptake classified as high or very high

Exclusion Criteria:

* Active smoker currently or within the past 5 years
* Regular intake of medication deemed by the responsible study physician to affect the test parameters (hormonal contraception is accepted for women)
* Chronic or acute illness deemed by the responsible study physician to affect the test parameters
* Deviation from the study protocol
* Lean mass index >21 kg/m²
* Pregnancy
* Smoker
* Blood donation during the past 3 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Urine concentration | Through study completion, an average on 1 week
  Difference in urine concentration with salmeterol administered before performance tests in different conditions

CONTACTS AND LOCATIONS:
Locations (1):
- August Krogh Building, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided